CLINICAL TRIAL: NCT06896890
Title: A Phase I/II First-in-human Trial Investigating Safety, Tolerability, Pharmacokinetics and Anti-tumour Activity of Ascending Doses of a Dry Powder Cisplatin Formulation for Inhalation to Treat Stage IV Non-small Cell Lung Cancer Patients
Brief Title: Cisplatin (CIS) Administered As Dry Powder for Inhalation (DPI) in Patients with Stage IV Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inhatarget Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIS-DPI-01
Record Dates: First submitted 2025-03-11; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: NSCLC (advanced Non-small Cell Lung Cancer); Stage IV Lung Cancer
Keywords: non-small cell lung cancer; NSCLC; cisplatin; inhaled; pulmonary administration route; CIS-DPI; Dry Powder for Inhalation; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Respiratory Aspiration | interventions — Inhalation

STUDY DESIGN:
Intervention Model Description: A Phase I/II First-in-Human Single-arm Open-label Multicentre Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cisplatin Dry Powder for Inhalation (CIS-DPI) (Experimental): Stage IV NSCLC patients with Programmed Death-Ligand Tumor Propensity Score (PDL1 TPS) ≥50% OR <50%, respectively receiving study treatment CIS-DPI combined with standard of care treatment (either iv pembrolizumab OR iv pembrolizumab and iv carboplatin-doublet chemotherapy (i.e. pemetrexed + carboplatin in non-squamous NSCLC patients or paclitaxel + carboplatin in squamous NSCLC patients)).
  Interventions: Drug: CIS-DPI

INTERVENTIONS:
Drug: CIS-DPI — * Administration of cisplatin by inhalation (pulmonary route) using single-use RS01 capsule-based device and CIS-DPI hard capsules containing 2.5 mg, 5 mg, and 10 mg cisplatin.
  * CIS-DPI, administered once-a-day, 5-days on followed by 2-days off. Daily dose to be administered will range from an initial dose of 2.5 mg cisplatin to a maximal theoretical dose of 30 mg (i.e., dose 1 to dose 7).
  Other Names: Cisplatin-based Dry Powder for Inhalation

SUMMARY:
The combination of chemotherapy and immunotherapy shows promising results in terms of overall survival (OS) and progression-free survival (PFS) for the treatment of first-line stage IV non-small cell lung cancer (NSCLC) patients, leading to such combinations becoming a real backbone of the Standard of Care (SoC) for NSCLC patients.

However, conventional chemotherapy's severe systemic toxicities represent a limiting factor in terms of administered dose and frequency. Administration of cisplatin by inhalation (pulmonary route) is a promising additional approach that may overcome the limitations of conventional chemotherapy.

Use of a dry powder inhaler enables a high therapeutic response by delivering high local concentrations of a well-established active substance without the usual undesired reactions that limit the use of high doses when administered through the conventional systemic route.

This study may provide insights into whether this add-on treatment might be a safe and potentially efficacious option for NSCLC patients.

DETAILED DESCRIPTION:
The survival of patients with metastatic lung cancer has significantly improved with platinum-based treatments and, more recently, with targeted therapies and immunotherapies. However, despite therapeutic advances, lung cancer remains the world's leading cause of cancer-related death (approximately 2 million per year), due to innate or acquired tumour resistance to treatments.

The combination of chemotherapy (platinum-doublets) and immunotherapy (immune checkpoint inhibitors) shows promising results in terms of overall survival (OS) and progression-free survival (PFS) for the treatment of first-line stage IV non-small cell lung cancer (NSCLC) patients, leading to such combinations becoming a real backbone of the Standard of Care (SoC) for NSCLC patients. These results may be attributable to the immunogenic effects of chemotherapy-induced tumour cell death, which, when used with immune checkpoint inhibitors, is an approach that may improve the clinical outcomes of cancer patients.

However, conventional chemotherapy's severe systemic toxicities represent a limiting factor in terms of administered dose and frequency, requiring long rest phases (i.e., interruption of treatment) leading to a relatively limited frequency of chemotherapy treatment in current clinical practice (4 to 6 cycles of intravenous (iv) administration, all separated by a 3-week interruption period). This limitation, associated with high mortality, especially in the advanced stages of lung cancer, demonstrates that the treatments/combinations currently used are far from optimal.

Administration of cisplatin by inhalation (pulmonary route) is a promising additional approach that may overcome the limitations of conventional chemotherapy and increase the efficacy of the current SoC via sustained local attack on the lung tumours of patients treated using immune checkpoint inhibitors with or without iv chemotherapy.

Use of a dry powder inhaler (DPI) enables a high therapeutic response by delivering high local concentrations of a well-established active substance without the usual undesired reactions that limit the use of high doses when administered through the conventional systemic route.

Thanks to limited systemic exposure to the cytotoxic active ingredient with the use of a dry powder inhaler, such add-on treatment enables considering 5 times weekly administration of inhaled chemotherapy at the patient's home. Increasing the frequency of local chemotherapy treatment in this way may enhance activation of the systemic anti-tumour immune response via local activation and stimulation of tumour-specific antigen release as a result of a safe, sustained and prolonged local effect, compared to the peak/short effect of iv chemotherapy.

This study may provide insights into whether this add-on treatment might be a safe option for NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥18 years of age at the time of signing the informed concent form (ICF).
* The patient must have a pathologically or cytologically confirmed Stage IV NSCLC that could be treated with pembrolizumab alone or combined with carboplatin/pemetrexed or paclitaxel.
* The patient must have measurable disease according to RECIST 1.1.
* The patient must be treatment naïve for stage IV NSCLC at the time of study enrolment. Patients having received, at least 6 months before D1, platinum derivatives adjuvant after (i) surgery or (ii) concomitant chemotherapy-radiotherapy for unresectable locally advanced NSCLC are eligible.
* The patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* The patient must have adequate organ function values as follows:

  1. Haematology:

     1. Platelet count >100,000 cells/mm3.
     2. Absolute neutrophil count >1,500 cells/mm3.
     3. Haemoglobin >9 g/dL.
  2. Serum creatinine less or equal to upper limit of normal (ULN) or creatinine clearance >60 mL/min/1.73 m2 on the basis of Cockcroft-Gault glomerular filtration rate estimation.
  3. Coagulation:

     1. International normalised ratio (INR) ≤1.5; for patients treated with coumarins INR ≤3 is acceptable.
     2. Prothrombin time (PTtest) and activated partial thromboplastin time (aPTT) <1.6 x ULN unless therapeutically warranted.
  4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3 x ULN. In case of hepatic metastasis, AST and ALT <5 x ULN.
  5. Bilirubin ≤1.5 x ULN, except for patients with known familial hyperbilirubinemia (such as Gilbert syndrome); for patients with documented Gilbert's syndrome (Gilbert-Meulengracht syndrome) total bilirubin of ≤3 x ULN is acceptable.
* The patient must have a resting oxygen saturation of at least 90%, a FEV1 ≥50% of predicted values as determined by spirometry and a DLCO of at least 50%.
* The patient is able to manipulate adequately the refillable single-dose (RS01) capsule-based device.
* Women of childbearing potential should have a negative serum pregnancy test, and be not pregnant or breastfeeding at screening.
* Male patients that are able to father children and female patients of childbearing potential must agree to use highly effective methods of contraception throughout the study and for at least 6 months after the last dose of CIS-DPI.
* The patient has given written informed consent prior to any study-specific procedures.
* The patient has the willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Patients with contraindication to or unwillingness to undergo contrast-enhanced computed tomography (CT) scans and chest X-rays according to the protocol requirements.
* Patients who are participating in an investigational drug or device study within 4 weeks prior to the planned day for the first study treatment administration (D1).
* Patients who have been treated by any anti-neoplastic agent within 6 months prior to the planned day for the first study treatment administration (D1).
* Patients who have received prior therapy with an immune checkpoint inhibitor.
* Patients who have received prior radiotherapy (head, neck, thorax, or abdomen) within 4 weeks prior to the planned day for the first study treatment administration (D1) except palliative radiotherapy (2 weeks). Patients must have recovered from all radiation-related toxicities, not require corticosteroids (see criterion 2425) and not have had radiation pneumonitis >grade 2.
* Patients with concurrent thoracic irradiation for the treatment of lung cancer.
* Patients who underwent major surgery within 4 weeks before the planned day for the first study treatment administration (D1).
* Patients with EGFR activating mutation or ALK translocation, or any other activable molecular alterations that in the opinion of the investigator could be more effectively treated with targeted therapies (Note: This exclusion criterion must be checked before the first SoC administration).
* Non-smoking patients without results of Epidermal growth factor receptor (EGFR) mutation and anaplastic large-cell lymphoma kinase (ALK) translocation before the planned day for the first study treatment administration (D1).
* Patients with known pre-existing hearing impairment due to VIII nerve alteration.
* Patients presenting a history of previous severe intolerance to or sensitivity to cisplatin, vitamin E or lactose.
* Patients with mouth problems (e.g. cleft palate) or other abnormalities that would prevent tight fit of the mouth seal.
* Patients with uncontrolled symptomatic pleural effusion or uncontrolled pneumothorax.
* Patients having undergone pneumonectomy or bilobectomy (except if bilobectomy includes the right middle lobe).
* Patients with a known history of severe cough/bronchospasm upon inhalation of dry powder inhalation products.
* Patients with a known history or current evidence of any chronic upper or lower respiratory conditions (other than asthma and allergic or non-allergic rhinitis). History of mild acute upper or lower respiratory conditions are allowed, provided that the condition has been resolved at least 3 months before the planned day for the first study treatment administration (D1) and provided that, in the investigator's judgement, this occurrence poses no additional risk for this subject.
* Patients with a known history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, acute exacerbation of chronic obstructive pulmonary disease (COPD) in the last 3 months before D1 (even if managed in an outpatient setting), known history of interstitial lung disease (ILD), or (non-infectious) pneumonitis that require steroids or that have current pneumonitis.
* Patients with uncontrolled asthma, as defined in the Global Initiative for Asthma (GINA) 2020 guidelines. Patients with (i) a history of asthma or (ii) controlled active asthma treated with long-acting beta-2 mimetics with or without inhaled corticosteroids and having less than one asthma crisis per month, are eligible.
* Patients with uncontrolled or severe active infection.
* Known positivity for human immunodeficiency virus (HIV) or history of HIV (HIV testing is not mandatory):
* Active hepatitis B virus (HBV; chronic or acute) defined as having a positive hepatitis B surface antigen (HBsAg) test at screening. Patients with past or resolved HBV infection (defined as having a negative HBsAg test and a positive hepatitis B core antigen antibody test) are eligible.
* Active hepatitis C virus (HCV) infection defined as having a positive HCV antibody test followed by a positive HCV ribonucleic acid (RNA) test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test. Patients who are positive for HCV antibodies are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
* Positivity for Coronavirus Disease 2019 (COVID-19) by PCR testing. PCR result must not be older than 72 hours prior to the planned day for the first study drug administration (D1). Completed vaccination or prior COVID-19 infection does not exempt patients from PCR testing.
* Live virus vaccine within 30 days prior to the planned day for the first study treatment administration (D1) (Note: inactivated seasonal flu vaccine is acceptable).
* Patients using oral corticosteroids within 4 weeks1 week prior to the planned day for the first study treatment administration (D1) above daily dose of 10 mg or any single dose of 16 mg. Patients receiving inhaled or topical corticosteroids are eligible.
* Patients who are presenting persistent toxicities greater than or equal to Common Terminology Criteria for Adverse Events (CTCAE version 5.0) grade 2 caused by previous cancer therapy (except for clinically non-significant toxicities, such as alopecia).
* Patients having a current active malignancy with the exception of adequately-treated basal or squamous cell carcinoma of the skin, preinvasive carcinoma of the cervix, in situ carcinoma of the breast or low-grade prostate cancer with no plan for treatment intervention. Patients with previous history of malignancy provided that patient has been free of disease for at least 3 years may be included.
* Patients with a known history of arterial thromboembolic event (ATE) or venous thromboembolic event (VTE) within 3 months prior to the planned day for the first study treatment administration (D1).
* Patients with a known history of any of the following conditions: presyncope or syncope of either unexplained or cardiovascular etiology, uncontrolled ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation) or sudden cardiac arrest.
* Patients with significant or uncontrolled congestive heart failure (CHF) with Left Ventricular Ejection Fraction Assessment (LVEF) of less than 40%, significant or uncontrolled myocardial infarction or significant ventricular arrhythmias within the last 6 months prior to the planned day for the first study treatment administration (D1).
* Patients who have uncontrolled hypertension defined as systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90 mmHg despite standard medical management with ≥2 anti-hypertensive drugs.
* Patients with a known history of organ transplant or current active immunosuppressive therapy (such as cyclosporine, tacrolimus).
* Patients with known history or presence of clinically relevant central nervous system (CNS) pathology, any autoimmune disease or significant coagulation disorder.
* Patients with carcinomatous meningitis or CNS metastases, except where such metastases are stable and already irradiated.
* Patients with peripheral neuropathy >grade 1.
* Patients with any significant medical condition that in the opinion of the investigator makes participation in the trial against the patients' best interests.
* Patients who are unwilling or unable to comply with the study protocol for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (dose escalation phase) | From first study treatment administration (Day 1) to the end of Week 12.
  Define the Maximum Tolerated Dose (MTD) based on Dose Limiting Toxicity (DLT). Dose-Limiting toxicity is defined to be a toxicity (i.e. confirmed investigational product related AE) that prevents further administration of the agent at that dose level.
Recommended Phase II dose (Safety expansion phase) | From the first study treatment administration (Day 1) to the end of Week 12.
  Confirm the recommended phase II dose (RP2D) based on Dose Limiting Toxicity (DLT). Dose-Limiting toxicity is defined to be a toxicity (i.e. confirmed investigational product related AE) that prevents further administration of the agent at that dose level.

SECONDARY OUTCOMES:
Pharmacodynamic markers | From first study treatment administration (Day 1) to the end of Week 12.
  To assess platinum plasma levels
CIS-DPI efficacy - Objective response rate (ORR) | From first study treatment administration (Day 1) to the end of Week 12.
  To assess the incidence of objective response (OR), stable disease (SD), progressive disease (DP) at each tumour response assessment planned according to the Response Evaluation Criteria in Solid Tumours version 1.1 (RECIST 1.1) and Immune Response Evaluation Criteria in Solid Tumours (iRECIST);
CIS-DPI efficacy - DCR | From first study treatment administration (Day 1) to the end of Week 12.
  To assess the disease control rate (DCR)
CIS-DPI efficacy - BOR | From first study treatment administration (Day 1) to the end of Week 12.
  To assess the best overall response (BOR);
CIS-DPI efficacy - DOR | From first study treatment administration (Day 1) to the end of Week 12.
  To assess the duration of response (DOR) for patients with OR;
CIS-DPI efficacy - OS | From first study treatment administration (Day 1) until the date of death from any cause, whichever came first, assessed up to 100 months
  To evaluate the Overall Survival (OS)
CIS-DPI efficacy - PFS | From first study treatment administration (Day 1) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  To evaluate the Progression Free survival (PFS).

OTHER OUTCOMES:
CIS-DPI induced Immune Reactions | From first study treatment administration (Day 1) to the end of Week 12.
  To assess cytokine levels.
CIS-DPI induced Immune Reactions | From first study treatment administration (Day 1) to the end of Week 12.
  To assess immune cell count.
CIS-DPI efficacy - RECIST 1.1 Tumor burden | From first study treatment administration (Day 1) to the end of Week 12.
  To assess tumour burden evolution using RECIST 1.1 analyses
CIS-DPI efficacy - iRECIST Tumor burden | From first study treatment administration (Day 1) to the end of Week 12.
  To assess tumour burden evolution using iRECIST analyses
CIS-DPI efficacy - volumetric Tumor burden | From first study treatment administration (Day 1) to the end of Week 12.
  To assess tumour burden evolution based on volumetric tumour load (VTL)
CIS-DPI efficacy CTM | From first study treatment administration (Day 1) to the end of Week 12.
  To assess circulating tumour markers (CTM)
CIS-DPI Safety | From first study treatment administration (Day 1) to the end of Week 12.
  To characterise and predict treatment safety based on quantitative imaging analysis extracted from computed tomography (CT) scans. To evaluate safety using quantitative imaging analysis features compared to the safety endpoints.
Pulmonary function parameters (PFT) - PIF | From first study treatment administration (Day 1) to the end of Week 12.
  Measure peak inspiratory flow (PIF)
Pulmonary function parameters (PFT) - PEF | From first study treatment administration (Day 1) to the end of Week 12.
  Measure peak expiratory flow (PEF)
Pulmonary function parameters (PFT) - FEV1 | From first study treatment administration (Day 1) to the end of Week 12.
  Measure forced expiratory volume in one second (FEV1)
Pulmonary function parameters (PFT) - FVC | From first study treatment administration (Day 1) to the end of Week 12.
  Measure forced vital capacity (FVC)
Pulmonary function parameters (PFT) - RV | From first study treatment administration (Day 1) to the end of Week 12.
  Measure residual volume (RV)
Pulmonary function parameters (PFT) - TLC | From first study treatment administration (Day 1) to the end of Week 12.
  Measure total lung capacity (TLC)
Pulmonary function parameters (PFT) - FRC | From first study treatment administration (Day 1) to the end of Week 12.
  Measure functional residual capacity (FRC)
Pulmonary function parameters (PFT) - DLCO | From first study treatment administration (Day 1) to the end of Week 12.
  Measure diffusing lung capacity for carbon monoxide (DLCO)
Pulmonary function parameters (PFT) - KCO | From first study treatment administration (Day 1) to the end of Week 12.
  Measure the carbon monoxide transfer coefficient (KCO)
Patient reported outcomes - Visual Analog Scale | From first study treatment administration (Day 1) to the end of Week 12.
  To collect before and within 30 minutes after CIS-DPI treatment a 10 point visual analog scale (the higher the better status) for general health status, cough, dyspnea, and throat irritation
CIS-DPI dose delivery | From first study treatment administration (Day 1) to the end of Week 12.
  To assay the cisplatin remaining in devices and capsules after use.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Berghmans, Prof.MD., Principal Investigator — Hopital Universitaire de Bruxelles (HUB)
Locations (15):
- Belgium (7):
  - Institut Jules Bordet - Hôpital Universitaire de Bruxelles, Brussels
  - GHDC, Charleroi
  - CHU Helora - Site Jolimont, Jolimont
  - AZ Groeninge, Kortrijk
  - CHU Sart Tilman, Liège
  - CHU Ambroise Paré, Mons
  - AZ Delta, Roeselare
- France (4):
  - Université Paris-Saclay, UVSQ, APHP - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Centre François Baclesse de Caen, Caen
  - Hôpital Européen Georges Pompidou, Paris-Cite University, Paris
  - L'Institut de Cancérologie de l'Ouest, Saint-Herblain
- Spain (4):
  - Instituto Oncologico Dr Rosell, Hospital Universitario Dexeus, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La PAZ, IdiPAZ, Madrid
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: Undecided